CLINICAL TRIAL: NCT02244476
Title: Validation Study to Evaluate the Use of Acoustic Tribology to Assess Mouthfeel of Dairy Drinks
Brief Title: Acoustic Tribology Validation Study
Status: Completed | Type: Observational
Sponsor: NIZO Food Research (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Other Study IDs: NIZO 105356
Record Dates: First submitted 2014-09-08; First posted 2014-09-19 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Mouth Feel in Relation to Food Preference and Energy Intake
Keywords: mouth feel; acoustic tribology; vibration spectrum; sensory perception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — tongue scrapings
Oversight: Data Monitoring Committee: No

SUMMARY:
Dairy-based beverages contain fat and sugars. As both contribute to the energy intake upon consumption, food industry strives to reduce these ingredients while maintaining the taste, texture and aroma properties of the beverages. A successful reduction of fat and sugar from drinks has still proven a great challenge since consumers have less preference for the mouth feel of reformulated beverages than for the regular beverages. Mainly because instrumental measures like rheology and traditional tribology do not entirely predict the experienced mouth feel, there is an interest in alternative correlates for mouth feel aspects related to fat and sugar perception. In a recent study it was demonstrated that vibrations produced during interaction between the tongue, palate and beverages during consumption are very sensitive to the amount of fat and texturizers in the beverage. The present study aims at clarifying that relation for a larger panel of human subjects, by systematically evaluating vibration spectra during consumption of dairy beverages that differ in fat content, sugar content or pH. Secondly, the correlation of vibration spectra (acoustic tribology) with mouth feel-related sensory properties and composition of fat deposits on the tongue will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Healthy set of teeth
* Ability to work with sensory descriptors for dairy products.
* Able to produce an acoustic signal that is larger than the background signal
* Voluntary participation
* Having given written informed consent
* Willing to comply with study procedures
* Willing to accept use of all encoded data, including publication, and the confidential use and storage of all data
* Willing to accept disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Wearing dentures
* Inability to comply with instructions for acoustic tribology
* A self-reported food allergy or sensitivity for ingredients of the test products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 16 volunteers from the local general population
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Powers in segments of time-frequency transferred vibration data | between 2s and 20s after consumption of each sip
  Spectral powers of acoustic signals (in V^2/s) produced by tongue-palate interactions during consumption of various foods in the bands 60-300Hz and 400-2000Hz.
Ratios of powers in segments of time-frequency transferred vibration data | 2-20 seconds after consumption of each sip
  Ratios of spectral powers in the 400-2000Hz band over powers in the 60-300Hz band of acoustic signals produced by tongue-palate interactions during consumption of various foods (unit-free).

SECONDARY OUTCOMES:
Reported rating of product thickness | 0-2 sec after consumption of each sip
  Evaluation of product thickness on a Visual Analogue Scale (mm distance from the lower anchor)
Relative fat content in the collected tongue coating | 2-20 sec after consumption of each sip
  percentage of fat encountered in tongue coating that was collected with a swab immediately after consumption
Reported rating of product Creaminess | 0-2 sec after consumption of each sip
  Evaluation of product creaminess on a Visual Analogue Scale (mm distance from the lower anchor)
Reported rating of product Roughness | 0-2 sec after consumption of each sip
  Evaluation of product roughness on a Visual Analogue Scale (mm distance from the lower anchor)
Relative sugar content in the collected tongue coating | 2-20 seconds after bite consumption
  percentage of sugars encountered in tongue coating that was collected with a swab immediately after consumption
Relative protein content in the collected tongue coating | 2-20 seconds after bite consumption
  percentage of protein encountered in tongue coating that was collected with a swab immediately after consumption

CONTACTS AND LOCATIONS:
Overall Officials: Harold Bult, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO food research, Ede, Netherlands